CLINICAL TRIAL: NCT06898255
Title: An Open-label, Multi-center, Phase I Study to Evaluate the Safety/Tolerability and Pharmacokinetics of GFS202A in Advanced Solid Tumor Patients With Pre-cachexia or Cachexia
Brief Title: A Phase I Study to Evaluate GFS202A in Advanced Solid Tumor Patients With Pre-cachexia or Cachexia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GFS202AX1101; CXSL2400937 (Other: NMPA)
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-03

CONDITIONS: Cancer Cachexia
Keywords: cachexia; cancer; GDF-15; IL-6
MeSH Terms: conditions — Cachexia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- GFS202A dose level 1 (Experimental)
  Interventions: Drug: GFS202A injection
- GFS202A dose level 2 (Experimental)
  Interventions: Drug: GFS202A injection
- GFS202A dose level 3 (Experimental)
  Interventions: Drug: GFS202A injection
- GFS202A dose level 4 (Experimental)
  Interventions: Drug: GFS202A injection
- GFS202A dose level 5 (Experimental)
  Interventions: Drug: GFS202A injection
- GFS202A dose level 6 (Experimental)
  Interventions: Drug: GFS202A injection

INTERVENTIONS:
Drug: GFS202A injection — Participants will receive GFS202A intravenously every 3 weeks (Q3W) in a 21-day cycle. The treatment duration was 12 weeks.

SUMMARY:
An open-label, multi-center, phase I study to evaluate the safety/tolerability and pharmacokinetics of GFS202A in advanced solid tumor patients with pre-cachexia or cachexia. The primary objective is to assess the safety/tolerability of GFS202A, determine its maximum tolerated dose (MTD), and recommend a dose range for future studies.

Enroll participants with cancer cachexia or precachexia to receive GFS202A monotherapy. During the study period, participants will undergo assessments for safety and preliminary efficacy according to the visit schedule. Pharmacokinetic, anti-drug antibody (ADA), and pharmacodynamic (PD) /biomarker samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and sign the informed consent form.
2. Men or women between the ages of 18 and 80 years at the time of written informed consent.
3. Patients with histologically or cytologically confirmed solid tumors. Pre-cachectic and cachectic patients with weight loss or baseline BMI < 21 kg/m2 within 6 months before the first study dose.
4. Persistent concomitant appetite/eating problems related to cancer.
5. It has adequate organ function.
6. The ECOG PS score was 0-2.
7. The investigator judged the expected survival time to be ≥ 3 months.

Exclusion Criteria:

1. With active brain metastases.
2. With other active diseases that lead to reduced food intake or seriously affect digestion and absorption
3. Baseline BMI > 28 kg/m2.
4. With infectious diseases.
5. With clinically significant cardiovascular disease.
6. With uncontrolled metabolic diseases.
7. With known clinically significant allergic reactions to antibodies and excipients.
8. With history of drug or alcohol abuse.
9. Pregnant or lactating female subjects or women planning to become pregnant during the study.
10. With pleural, peritoneal, or pericardial effusion that causes overt symptoms or requires repeated drainage (frequency ≥ 1 time/month).
11. Use of any investigational drug within 28 days before the first study dose or within five half-lives of the drug, whichever was shorter, or planned for the duration of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE/SAE | Up to 6 weeks after the last dose
Incidence of DLT | Up to 21 days after the first dose

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Baseline, up to 6 weeks after the last dose
Area under the plasma concentration versus time curve (AUC) | Baseline, up to 6 weeks after the last dose
Trough Plasma Concentration (Ctrough) | Baseline, up to 6 weeks after the last dose
Half-life (T1/2) | Baseline, up to 6 weeks after the last dose
Incidence of ADA | Baseline, up to 6 weeks after the last dose
Concentration of GDF-15 and IL-6 | Baseline, up to 6 weeks after the last dose
Weight change from baseline | Baseline, up to 6 weeks after the last dose
L3SMI change from baseline | Baseline, up to 6 weeks after the last dose
Change from baseline in Functional Assessment of Anorexia-Cachexia Therapy (FAACT-ACS) scores | Baseline, up to 6 weeks after the last dose
Change from baseline in Functional Assessment of Cancer Therapy-General (FACT-G) scores | Baseline, up to 6 weeks after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun-Yat Sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No